CLINICAL TRIAL: NCT00111579
Title: A Prospective, Randomized, Open-Label Study to Evaluate the Immune Responses of Trivalent Cold-Adapted Influenza Vaccine (CAIV-T) Compared With Trivalent Inactivated Vaccine (TIV) in Children 6 to <36 Months of Age
Brief Title: Study to Evaluate the Immune Responses of Trivalent Cold-Adapted Influenza Vaccine (CAIV-T) Compared With (TIV)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Chris Ambrose, Dir. Medical Affairs, MedImmune LLC
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP123
Record Dates: First submitted 2005-05-23; First posted 2005-05-24 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2008-07

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — FluMist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): CAIV-T
  Interventions: Biological: CAIV-T
- 2 (Other): TIV
  Interventions: Other: TIV

INTERVENTIONS:
Biological: CAIV-T — A total vol. of 0.2 mL will be administered intranasally (approx. 0.1 mL into each nostril)for ea. of two doses.
  Arms: 1
Other: TIV — A total vol. of 0.25 will be administered intramuscularly for each of two doeses.
  Arms: 2

SUMMARY:
The purpose of this study is to describe the level of serum antibody conferred by CAIV-T and TIV against homotypic and heterotypic influenza virus strains.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Ages 6 to but less than 36 months (reached their 6th month but have not yet reached their 3rd birthday) at the time of randomization
* Written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization (if applicable) obtained from the participant's parent/legal representative
* Ability of the parent/legal representative to understand and comply with the requirements of the study
* Parent/legal representative available by telephone
* Ability to complete follow-up period of 180 days after final study vaccination, as required by the protocol

Exclusion Criteria:

* History of hypersensitivity to any component of CAIV-T or TIV, including egg or egg products, monosodium glutamate, porcine gelatin or thimerosal
* History of hypersensitivity to gentamicin
* Any known immunosuppressive condition or immune deficiency disease (including HIV infection), or ongoing receipt of any immunosuppressive therapy
* Household contact who is immunocompromised (participants should also avoid close contact with immunocompromised individuals for at least 21 days after each study vaccination)
* History of Guillain-Barre syndrome
* Medically diagnosed wheezing, bronchodilator use, or steroid use (systemic or inhaled), by parent/legal representative report or chart review, within the 42 days prior to randomization (i.e., children with recent persistent asthma are excluded); or history of severe persistent asthma, according to the criteria described in the National Asthma Education and Prevention Program (NAEPP) Expert Panel Report: Guidelines for the Diagnosis and Management of Asthma - Update on Selected Topics 2002
* Acute febrile (not greater than 100.0 degrees F oral or equivalent) and/or clinically significant respiratory illness (e.g., cough or sore throat) within 72 hours prior to either study vaccination
* Use of aspirin or aspirin-containing products within 30 days prior to randomization, or expected use through 180 days after final study vaccination
* Receipt of any prior influenza vaccine
* Use of anti-influenza medications (including amantadine, rimantadine, oseltamivir, and zanamivir) within 14 days prior to randomization, or expected use through 180 days after final study vaccination
* Administration of any live virus vaccine within 30 days prior to randomization, or expected receipt through 30 days after final study vaccination
* Administration of any inactivated (i.e., non-live) vaccine within 14 days prior to randomization, or expected receipt within 14 days before, or 14 days after, either study vaccination
* Receipt of any investigational agent within 30 days prior to randomization, or expected receipt through 180 days after final study vaccination (use of licensed agents for indications not listed in the package insert is permitted)
* Receipt of any blood product within 90 days prior to randomization, or expected receipt through 180 days after final study vaccination
* Family member or household contact who is an employee of the research center or otherwise involved with the conduct of the study
* Any condition that, in the opinion of the investigator, would interfere with evaluation of the vaccine or interpretation of the study results

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52
Dates: Start 2005-05; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
The following immunogenicity endpoints: The strain-specific HAI seroconversion rates (≥ 4-fold increase) among baseline seronegative participants (HAI titer ≤ 1:4), by dose number | Day 28 post final vaccination
The proportion of participants achieving ≥ 4-fold increase in strain-specific HAI titer from baseline in all participants regardless of baseline serostatus, by dose number | Day 28 post final vaccination

SECONDARY OUTCOMES:
Safety endpoints include: AEs SAEs and significant new medical conditions for all participants | Day 28 post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Robert Walker, MD, Study Director — MedImmune LLC
Locations (5):
- United States (5):
  - Wee Care Pediatrics, Layton, Utah
  - Bear Care Pediatrics, Ogden, Utah
  - Alpine Pediatrics, Pleasant Grove, Utah
  - Utah Valley Pediatrics, Provo, Utah
  - Families First Pediatrics, South Jordan, Utah